CLINICAL TRIAL: NCT06468735
Title: The Relationship Among Sarcopenia, Preperitoneal Fat Thickness and Cholecystectomy: The Good, The Bad and The Ugly
Brief Title: The Relationship Among Sarcopenia, Preperitoneal Fat Thickness and Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semih Sezer, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CholecystectomySarcopenia
Record Dates: First submitted 2024-06-19; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sarcopenia; Cholecystectomy
Keywords: ultrasound; Quadriceps; gall bladder; IsarcoPRM
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cholecystectomy (Experimental): Ultrasonography-guided assessment of sarcopenia and measurement of visceral, preperitoneal, subcutaneous maximum and subcutaneous minimum fat thickness in cholecystectomised participants
  Interventions: Diagnostic Test: sarcopenia assessment; Diagnostic Test: visceral fat thickness measurement
- Control (Experimental): Ultrasonography-guided assessment of sarcopenia and measurement of visceral, preperitoneal, subcutaneous maximum and subcutaneous minimum fat thickness in participants without cholecystectomy
  Interventions: Diagnostic Test: sarcopenia assessment; Diagnostic Test: visceral fat thickness measurement

INTERVENTIONS:
Diagnostic Test: sarcopenia assessment — Quadriceps muscle thickness measurement at the midpoint between the anterior superior iliac spine and the upper pole of the patella.
  Sarcopenia assessment The quadriceps muscle thickness (mm) was divided by the BMI to get the sonographic thigh adjustment ratio (STAR) values. Grip strength was assessed using an electronic hand dynamometer on the dominant hand side. Three measurements were obtained from the dominant hand and the maximum value was taken for the analyses. Participants in the chair stand test (CST) were instructed to rapidly rise and fall from a chair five times while keeping their arms folded across their chests. The test was repeated three times, and the mean time was recorded. Together with low STAR values (<1.0 for females and <1.4 for males), having low grip strength (<19 kg for females or <32 kg for males) and/or prolonged CST duration (≥12 seconds) were used to diagnose sarcopenia
Diagnostic Test: visceral fat thickness measurement — Intraabdominal visceral adipose tissue thickness was calculated by placing the probe 2-cm proximal to the midline of the umbilicus with minimal pressure and measuring the distance from the inner surface of the linea alba to the anterior wall of the abdominal aorta. Subcutaneous maximum fat thickness was measured from the distance between the subcutaneous tissue and the linea alba from the same point. Preperitoneal fat thickness was measured from the distal neighborhood of the xiphoid process, 1.5 cm to the right side of the widest distance between the parietal peritoneum and the linea alba. Minimum subcutaneous fat thickness was calculated as the distance measured from the distal neighborhood of the xiphoid process, measured as the shortest distance between the outer part of the linea alba and the subcutaneous fat tissue.

SUMMARY:
The aim of this study was to examine the relationship between sarcopenia and visceral adiposity in participants with and without cholecystectomy.

In this way, the long-term effects of cholecystectomy operations, which are commonly performed in the society and thought to be harmless, will be evaluated.

DETAILED DESCRIPTION:
Cholecystectomy is recognized as a harmless operation with low mortality and morbidity and is commonly performed worldwide. The unexplained increase in metabolic disorders such as dyslipidemia, hyperglycemia, non-alcoholic fatty liver disease (NAFLD) and sarcopenia with cholecystectomy in recent studies has led to the need for further investigation of these patients. There are very few studies investigating the relationship among sarcopenia, visceral adiposity and cholecystectomy. In previous studies, BIA or DEXA was used for sarcopenia assessment and non-US methods were used for visceral fat assessment. In our study, we aimed to determine the relationship among sarcopenia, visceral adipose tissue and cholecystectomy by using US, which is an easy, cheap and a valid/reliable method.

A total of 158 community-dwelling patients (aged between 41 to 80 years), including cholecystectomized (N=89) and non-cholecystectomized (N=69) participants from gastroenterology clinics were included.

Sarcopenia assessment The quadriceps muscle thickness (mm) was divided by the BMI to get the sonographic thigh adjustment ratio (STAR) values. Grip strength was assessed using an electronic hand dynamometer on the dominant hand side. Three measurements were obtained from the dominant hand and the maximum value was taken for the analyses. Participants in the chair stand test (CST) were instructed to rapidly rise and fall from a chair five times while keeping their arms folded across their chests. The test was repeated three times, and the mean time was recorded. Together with low STAR values (<1.0 for females and <1.4 for males), having low grip strength (<19 kg for females or <32 kg for males) and/or prolonged CST duration (≥12 seconds) were used to diagnose sarcopenia.

Intraabdominal visceral adipose tissue thickness was calculated by placing the probe 2-cm proximal to the midline of the umbilicus with minimal pressure and measuring the distance from the inner surface of the linea alba to the anterior wall of the abdominal aorta. Subcutaneous maximum fat thickness was measured from the distance between the subcutaneous tissue and the linea alba from the same point. Preperitoneal fat thickness was measured from the distal neighborhood of the xiphoid process, 1.5 cm to the right side of the widest distance between the parietal peritoneum and the linea alba. Minimum subcutaneous fat thickness was calculated as the distance measured from the distal neighborhood of the xiphoid process, measured as the shortest distance between the outer part of the linea alba and the subcutaneous fat tissue.

ELIGIBILITY:
Inclusion Criteria:

* Cholecystectomy at least 5 years ago
* control group; those without cholecystectomy

Exclusion Criteria:

* Advanced cardiac, hepatic and renal insufficiency,
* active malignancies (currently or within the last one year receiving radiotherapy/chemotherapy),
* rheumatological diseases,
* severe knee, hip and hand osteoarthritis,
* use of any assistive device for walking,
* neuromuscular diseases (motor neuron diseases, polyneuropathies, myasthenia gravis),
* major depression,
* Parkinson's disease, previous stroke, cerebellar diseases and multiple sclerosis were excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
STAR values | through study completion, an average of 4 months
  <1.0 for females and <1.4 for males Quadriceps thickness(mm) /BMI kg/m2
low grip strength | through study completion, an average of 4 months
  <19 kg for females or <32 kg for males
chair stand test duration | through study completion, an average of 4 months
  ≥12 seconds
visceral adipose tissue thickness | through study completion, an average of 4 months
  mm
Subcutaneous maximum fat thickness | through study completion, an average of 4 months
  mm
Subcutaneous minimum fat thickness | through study completion, an average of 4 months
  mm
Preperitoneal fat thickness | through study completion, an average of 4 months
  mm

SECONDARY OUTCOMES:
BMI | through study completion, an average of 4 months
  kg/m2
Waist circumference | through study completion, an average of 4 months
  cm

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)